CLINICAL TRIAL: NCT04854421
Title: Evaluation of the Accuracy of a Computer Vision-based Tool for Assessment of Total Body Fat Percentage
Acronym: MEASURE
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Amazon, Inc. (Industry); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven Heymsfield, Professor, George A. Gray Endowed Chair, Pennington Biomedical Research Center
Other Study IDs: PBRC 2020-012
Record Dates: First submitted 2021-04-18; First posted 2021-04-22 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy adults: Community dwelling and have no life-threatening conditions or diseases that would alter body composition from what is typical for their age, sex, ethnicity, and BMI.
  Interventions: Device: VBC

INTERVENTIONS:
Device: VBC — Body Composition will be measured using the VBC system that takes under 60 seconds per scan. Image capture for VBC will include taking a series of four photos using a smartphone camera. Data from the camera will be downloaded to a local computer and then securely sent to the cloud for automated analysis and results generation. We will conduct two consecutive scans (image captures) for each research participant.

SUMMARY:
This research study is designed to validate the precision and accuracy of body measurement and composition results from a novel 2D imaging device that operates through a smart-phone application. Measurement references will be obtained through dual energy x-ray absorptiometry, air displacement plethysmography, bioelectrical impedance analysis, manual anthropometry, and previously validated 3D optical scanners.

DETAILED DESCRIPTION:
Participation in this study will require a single 3-hour visit to complete. Each person will be asked to arrive at PBRC wearing easily removable gym-style clothing. Upon checking in, they will first complete the informed consent process, then have their vital signs checked, and then women of child-bearing potential will also have a urine sample taken. Outpatient clinic procedures will be followed by a series of body size and composition assessments that will require an outfit of minimal clothing. Clean spandex shorts, sports bras, and lycra caps will be provided.

* Anthropometric measurements including hip, waist, arms, and thighs circumferences will be collected by a trained observer using a calibrated tape measure.
* Body shape will be measured digitally using 2D and 3D optical devices that optimize light patterns to calculate depth.
* Bioelectrical Impedance Analysis measures the amount of fat and lean mass in the body using electrodes positioned close to the feet and hands.
* Whole body dual-energy X-ray absorptiometry measures the amount of bone, muscle, and fat mass in the body using low energy X-rays.
* Air displacement plethysmography estimates whole body volume, fat mass, and fat-free mass of the body using variations in air pressure

ELIGIBILITY:
Inclusion Criteria:

* Being either male or female
* Being from 21 to 80 years of age
* Having a body weight of less than 440 pounds
* Being willing to comply with the study procedures

Exclusion Criteria:

* Being pregnant or attempting to become pregnant
* Having medical implants such as a pacemaker or metal joint replacements
* Having undergone any previous body altering procedures such as breast augmentation or amputation
* Having a body weight greater than 440 pounds

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants will be community dwelling and have no life-threatening conditions or diseases that would alter their body composition from what is typical for their age, sex, ethnicity, and BMI. Overall, participants must be ambulatory, able to withstand lying flat on the DXA table for up to 10 minutes, stand without aid for 2 minutes, weigh less than 440 lbs and be of generally good health.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Heymsfield, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (2):
- United States (2):
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Majmudar MD, Chandra S, Yakkala K, Kennedy S, Agrawal A, Sippel M, Ramu P, Chaudhri A, Smith B, Criminisi A, Heymsfield SB, Stanford FC. Smartphone camera based assessment of adiposity: a validation study. NPJ Digit Med. 2022 Jun 29;5(1):79. doi: 10.1038/s41746-022-00628-3. PMID 35768575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8/12/2020 through 10/21/2020 to undergo body composition assessments at one of two locations, Pennington Biomedical Research Center (PBRC) in Baton Rouge, Louisiana or the Weight Center of Massachusetts General Hospital (MGH) in Boston Massachusetts. Participants assessed at PBRC were recruited from the surrounding community using advertisements promoted by the facility's Recruitment Department. Those assessed at MGH were ongoing patients seen at the center.
Groups:
- Male Participants; Female Participants: Community dwelling and have no life-threatening conditions or diseases that would alter body composition from what is typical for their age, sex, ethnicity, and BMI.
Period: Overall Study
Arm/Group | Male Participants | Female Participants
Started | 54 | 84
Completed | 52 | 82
Not Completed | 2 | 2
Not completed — Removed from the final analysis due to poor image quality. | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Male Participants | Female Participants | Total
Number analyzed (Participants) | 52 | 82 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.1 (14.4) | 43 (14.8) | 43 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 82 | 82
  Male | 52 | 0 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 47 | 76 | 123
  Unknown or Not Reported | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 21 | 32
  White | 31 | 50 | 81
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 3 | 4 | 7
Height [Mean (Standard Deviation); unit: Centimeters] | 175.6 (8.7) | 163.0 (7.6) | 167.8 (10.2)
Weight [Mean (Standard Deviation); unit: Kilograms] | 92.8 (19.7) | 78.3 (19.4) | 84.0 (20.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter] | 30.0 (5.6) | 29.5 (7.0) | 29.7 (6.5)
Waist Circumference [Mean (Standard Deviation); unit: Centimeters] | 102.2 (14.3) | 92.2 (16.3) | 98.5 (15.7)
Hip Circumference [Mean (Standard Deviation); unit: Centimeters] | 108.2 (11.5) | 110.1 (14.3) | 109.4 (13.2)
Waist-to-hip Ratio [Mean (Standard Deviation); unit: Ratio] | 0.94 (0.08) | 0.87 (0.07) | 0.90 (0.08)
DXA %BF [Mean (Standard Deviation); unit: Percentage] — Dual-Energy X-ray Absorptiometry (DXA) percentage of total body fat
  Percentage | 28.6 (6.4) | 39.4 (7.2) | 35.2 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Body Fat Percentage Estimates to DXA References Classified by Body Mass Index
Description: Comparison of Body Fat Percentage estimates to DXA references classified by Body Mass Index
Time Frame: within a single, 3-hour evaluation
Population: A total of 406 adults were screened for this study. Of those,199 met all inclusion and exclusion criteria and were considered eligible. 138 participants were enrolled into the clinical study and 134 participants (64 from MGH and 70 from PBRC) were included in the final analysis; four participants (2.9%) were removed from the final analysis due to poor image quality. Participants at PBRC underwent ADP (N = 70). Note that DXA images were never used, only their derived Body Fat percentage.
Measure: Mean (Standard Deviation); unit: Total Body Fat Percentage
Groups:
- Smartphone Visual Body Composition (VBC): VBC: Body Composition was measured using the VBC system that takes under 60 seconds per scan. Image captured for VBC included taking a series of four photos using a smartphone camera.
- FitBit Aria 2 (cBIA 1); Tanita BF-684W (cBIA 2); Renpho ES-24M-W/B (cBIA 3): Three consumer weight scales capable of BIA-based body composition analysis were included in the protocol: FitBit Aria 2 (Fitbit, San Francisco, CA); Tanita BF-684W (Tanita, Tokyo, Japan); and Renpho ES-24M-W/B (Joicom Corporation, Anaheim, CA). These scales are designated as cBIA 1, cBIA 2, and cBIA 3.(Consumer Bio-Impedance Analysis)
- InBody S10 (pBIA1); Quantum IV (pBIA 2): All participants also underwent professional BIA (pBIA) at PBRC with an InBody S10 (InBody Co., Seoul, Korea) and at MGH with a RJL system (Quantum IV, RJL Systems, Clinton Township, MI, USA.). The RJL system uses a single frequency (50 Khz) and four gel adhesive electrodes. Instead, InBody is multi-frequency and uses contact electrodes. InBody and RJL are designated as pBIA1 and pBIA 2, respectively, in the sections that follow and were analyzed separately. (Professional Bio-Impedance Analysis).
- BOD POD ADP: Participants who were evaluated at PBRC (N = 70) also had %BF assessed with the BOD POD Air displacement plethysmography (ADP) device (BodPod Gold Standard Body Composition Tracking System, COSMED, Rome, Italy).
Arm/Group | Smartphone Visual Body Composition (VBC) | FitBit Aria 2 (cBIA 1) | Tanita BF-684W (cBIA 2) | Renpho ES-24M-W/B (cBIA 3) | InBody S10 (pBIA1) | Quantum IV (pBIA 2) | BOD POD ADP
Number analyzed (Participants) | 134 | 123 | 131 | 131 | 70 | 64 | 70
Total Body Fat Percentage
  BMI < 25: number analyzed (Participants) | 34 | 32 | 33 | 34 | 23 | 11 | 23
  BMI < 25 | 2.50 (1.8) | 6.36 (3.5) | 5.75 (3.3) | 7.66 (4.6) | 4.29 (2.2) | 4.41 (2.8) | 3.31 (2.2)
  BMI 25-29.9: number analyzed (Participants) | 45 | 40 | 43 | 43 | 21 | 24 | 21
  BMI 25-29.9 | 1.90 (1.4) | 3.02 (2.3) | 5.04 (14.3) | 6.00 (4.9) | 2.49 (1.4) | 3.82 (3.1) | 2.30 (1.9)
  BMI > 30: number analyzed (Participants) | 55 | 51 | 55 | 54 | 26 | 29 | 26
  BMI > 30 | 2.16 (1.4) | 4.44 (1.8) | 4.31 (3.6) | 4.60 (4.6) | 2.63 (2.0) | 5.58 (2.6) | 3.67 (2.3)

2. Primary Outcome: Comparison of Body Fat Percentage Estimates to DXA References Classified by Sex
Description: Comparison of Body Fat Percentage estimates to DXA references classified by Sex
Time Frame: within a single, 3-hour evaluation
Population: total of 406 adults were screened for this study. Of those,199 met all inclusion and exclusion criteria and were considered eligible. 138 participants were enrolled into the clinical study and 134 participants (64 from MGH and 70 from PBRC) were included in the final analysis; four participants (2.9%) were removed from the final analysis due to poor image quality. Participants at PBRC underwent ADP (N = 70). Note that DXA images were never used, only their derived Body Fat percentage.
Measure: Mean (Standard Deviation); unit: Total Body Fat Percentage
Arm/Group | Smartphone Visual Body Composition (VBC) | FitBit Aria 2 (cBIA 1) | Tanita BF-684W (cBIA 2) | Renpho ES-24M-W/B (cBIA 3) | InBody S10 (pBIA1) | Quantum IV (pBIA 2) | BOD POD ADP
Number analyzed (Participants) | 134 | 123 | 131 | 131 | 70 | 64 | 70
Total Body Fat Percentage
  Male Participants: number analyzed (Participants) | 52 | 46 | 50 | 49 | 27 | 25 | 27
  Male Participants | 1.88 (1.3) | 4.53 (5.0) | 6.23 (13.4) | 4.11 (3.3) | 3.37 (2.4) | 5.01 (3.0) | 3.50 (2.4)
  Female Participants: number analyzed (Participants) | 82 | 77 | 81 | 82 | 43 | 39 | 43
  Female Participants | 2.34 (1.6) | 4.45 (3.3) | 4.10 (3.1) | 6.89 (5.3) | 2.98 (1.8) | 4.54 (2.9) | 2.90 (2.1)

ADVERSE EVENTS:
Time Frame: Participants were monitored over the course of a single 4-hour visit to the facility.
Description: This was a minimal risk study. The VBC device consists of an external camera that is no more dangerous to a participant that taking his/her picture using a cellular device.
Groups:
- Male Participants; Female Participants: Community dwelling and have no life-threatening conditions or diseases that would alter body composition from what is typical for their age, sex, ethnicity, and BMI.
  VBC: Body Composition will be measured using the VBC system that takes under 60 seconds per scan. Image capture for VBC will include taking a series of four photos using a smartphone camera. Data from the camera will be downloaded to a local computer and then securely sent to the cloud for automated analysis and results generation. We will conduct two consecutive scans (image captures) for each research participant.
Arm/Group | Male Participants | Female Participants
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/82
Other Adverse Events (participants affected / at risk) | 0/52 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/21/NCT04854421/Prot_SAP_002.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/21/NCT04854421/ICF_003.pdf